CLINICAL TRIAL: NCT00321373
Title: A Study to Demonstrate the Non-Inferiority of Influenza Vaccine Candidate, Compared With Fluarix™ Administered Intramuscularly in Elderly Aged 60 Years Old and Above
Brief Title: Study to Evaluate an Influenza Vaccine Candidate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 107022; 107191 (Other: GSK)
Record Dates: First submitted 2006-03-16; First posted 2006-05-03 (Estimated); Results first posted 2013-05-01 (Estimated); Last update posted 2018-06-08 (Actual); Status verified 2016-09

CONDITIONS: Influenza
Keywords: Influenza; Influenza vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- GSK1247446A-AS03 Group (Experimental): Subjects aged 60 years or older at the time of the vaccination who received 1 dose of GSK1247446A vaccine adjuvanted with AS03. The vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: Candidate Influenza Vaccine GSK1247446A - 2 different formulations
- GSK1247446A Group (Experimental): Subjects aged 60 years or older at the time of the vaccination who received 1 dose of non-adjuvanted GSK1247446A vaccine. The vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: Candidate Influenza Vaccine GSK1247446A - 2 different formulations
- Fluarix Group (Active Comparator): Subjects aged 60 years or older at the time of the vaccination who received 1 dose of Fluarix vaccine. The vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: FluarixTM

INTERVENTIONS:
Biological: Candidate Influenza Vaccine GSK1247446A - 2 different formulations — Single dose, Intramuscular injection
  Arms: GSK1247446A Group; GSK1247446A-AS03 Group
Biological: FluarixTM — Single dose, Intramuscular injection
  Arms: Fluarix Group

SUMMARY:
The purpose of this study is to evaluate the immune response and safety of influenza vaccine candidate with or without adjuvant compared to Fluarix™ administered intramuscularly in elderly aged 60 years old and above.

DETAILED DESCRIPTION:
Subjects will be randomized into 3 groups and will be followed for 6 months with 4 scheduled contacts per subjects. The immune response will be evaluated at days 0, 21 and 180 after vaccination. The safety evaluation will involve follow-up of solicited local and general signs and symptoms, unsolicited adverse events and serious adverse events.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion criteria:

* A male or female age 60 years or older at the time of the vaccination.
* Subjects who the investigator believes can and will comply with the requirements of the protocol
* Written informed consent obtained from the subject.
* Free of an acute aggravation of the health status as established by clinical examination before entering into the study.

Exclusion criteria:

* Use of any investigational or non-registered product (drug or vaccine) within 30 days preceding the administration of the study vaccine, or planned use during the study period.
* Acute clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within three months prior to the first vaccine dose.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the first dose of study vaccine or planned administration during the study period.
* Administration of other licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to enrolment in this study. Planned administration of a vaccine not foreseen by the study protocol up to 30 days after vaccination.
* History of hypersensivity to a previous dose of influenza vaccine.
* Previous vaccination against influenza within the 9 months prior to enrollment.
* History of confirmed influenza infection within the last 12 months.
* History of allergy or reactions likely to be exacerbated by any component of the vaccine(s)
* Acute disease at the time of enrolment.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1220 (Actual)
Dates: Start 2006-05-11; Primary Completion 2006-07-01 (Actual); Study Completion 2006-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (15):
- Finland (9):
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Jarvenpaa
  - GSK Investigational Site, Kotka
  - GSK Investigational Site, Lahti
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Pori
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
  - GSK Investigational Site, Vantaa
- Greece (6):
  - GSK Investigational Site, Goudi / Athens
  - GSK Investigational Site, Haidari
  - GSK Investigational Site, Marousi
  - GSK Investigational Site, Nikaia Piraeus
  - GSK Investigational Site, Orestiáda
  - GSK Investigational Site, Thessaloniki

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 107022 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 107022 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 107022 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 107022 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 107022 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1220 subjects were enrolled in the study. Study duration was of approximately 6 months (180 days) for all subjects.
Period: Overall Study
Arm/Group | GSK1247446A-AS03 Group | GSK1247446A Group | Fluarix Group
Started | 407 | 406 | 407
Completed | 405 | 406 | 404
Not Completed | 2 | 0 | 3
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Other | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK1247446A-AS03 Group | GSK1247446A Group | Fluarix Group | Total
Number analyzed (Participants) | 407 | 406 | 407 | 1220
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.0 (5.12) | 64.1 (4.95) | 64.2 (5.38) | 64.1 (5.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 209 | 205 | 208 | 622
  Male | 198 | 201 | 199 | 598

OUTCOME MEASURES:

1. Primary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against 3 Strains of Influenza Virus
Description: Titers are presented as geometric mean titers (GMTs). The 3 flu strains assessed were A/New Caledonia, A/New York and B/Malaysia. The reference seropositivity cut-off value was ≥ 1:10.
Time Frame: At Days 0 and 21 post-vaccination
Population: The analysis was based on the ATP cohort for immunogenicity at Day 21 including subjects for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination at this time point.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | GSK1247446A-AS03 Group | GSK1247446A Group | Fluarix Group
Number analyzed (Participants) | 395 | 393 | 389
titer
  A/New Caledonia, Day 0 [N=395,393,389] | 13.4 [12.3 to 14.8] | 13.9 [12.6 to 15.3] | 14.2 [13.0 to 15.6]
  A/New York, Day 0 [N=395,393,389] | 10.8 [9.9 to 11.8] | 11.9 [10.7 to 13.1] | 11.5 [10.5 to 12.7]
  B/Malaysia, Day 0 [N=395,393,389] | 17.8 [16.0 to 19.7] | 16.0 [14.4 to 17.8] | 15.6 [14.0 to 17.4]
  A/New Caledonia, Day 21 [N=395,393,389] | 168.0 [148.5 to 190.1] | 97.7 [85.7 to 111.3] | 202.4 [177.4 to 230.9]
  A/New York, Day 21 [N=395,393,389] | 179.8 [159.3 to 202.9] | 70.4 [61.3 to 80.7] | 104.3 [91.5 to 118.9]
  B/Malaysia, Day 21 [N=394,390,389] | 341.2 [305.7 to 380.9] | 175.4 [154.1 to 199.5] | 292.0 [257.1 to 331.5]

2. Secondary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against 3 Strains of Influenza Virus
Description: as for outcome 1
Time Frame: At Day 180 post-vaccination.
Population: The analysis was based on the ATP cohort for immunogenicity at Day 180 including subjects for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination at this time point.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | GSK1247446A-AS03 Group | GSK1247446A Group | Fluarix Group
Number analyzed (Participants) | 389 | 383 | 380
titer
  A/New Caledonia at Day180 | 64.3 [57.6 to 71.8] | 54.3 [48.3 to 61.0] | 84.4 [74.8 to 95.3]
  A/New York at Day180 | 56.8 [50.9 to 63.5] | 35.8 [31.7 to 40.3] | 42.4 [37.7 to 47.6]
  B/Malaysia at Day180 | 88.6 [79.0 to 99.3] | 65.2 [58.0 to 73.3] | 90.9 [80.7 to 102.5]

3. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms.
Description: Assessed solicited local symptoms were ecchymosis, pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 ecchymosis/redness/swelling = ecchymosis/redness/swelling spreading beyond 50 millimeters (mm) of injection site.
Time Frame: During the 7-day (Days 0-6) follow-up period after vaccination
Population: The analysis was based on the Total Vaccinated Cohort that included all vaccinated subjects with the symptom sheet completed.
Measure: Number; unit: Subjects
Arm/Group | GSK1247446A-AS03 Group | GSK1247446A Group | Fluarix Group
Number analyzed (Participants) | 405 | 404 | 406
Subjects
  Any Pain | 246 | 32 | 86
  Grade 3 Pain | 12 | 0 | 1
  Any Ecchymosis | 28 | 20 | 19
  Ecchymosis > 50mm | 1 | 0 | 1
  Any Redness | 95 | 50 | 65
  Redness > 50mm | 22 | 1 | 6
  Any Swelling | 84 | 8 | 50
  Swelling > 50mm | 19 | 0 | 4

4. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms.
Description: Assessed solicited general symptoms were arthralgia, fatigue, fever [defined as oral temperature equal to or above 37.5 degrees Celsius (°C)], headache, muscle aches, shivering. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 7-day (Days 0-6) follow up period after vaccination
Population: The analysis was based on the Total vaccinated Cohort which included all vaccinated subjects with the symptom sheet completed.
Measure: Number; unit: Subjects
Arm/Group | GSK1247446A-AS03 Group | GSK1247446A Group | Fluarix Group
Number analyzed (Participants) | 405 | 404 | 406
Subjects
  Any Arthralgia | 80 | 17 | 21
  Grade 3 Arthralgia | 6 | 0 | 1
  Related Arthralgia | 73 | 14 | 18
  Any Fatigue | 149 | 42 | 47
  Grade 3 Fatigue | 6 | 1 | 0
  Related Fatigue | 148 | 36 | 42
  Fever (oral) ≥37.5°C | 21 | 4 | 2
  Fever (oral) ≥39.0°C | 0 | 0 | 0
  Related Fever | 21 | 2 | 1
  Any Headache | 104 | 51 | 53
  Grade 3 Headache | 5 | 0 | 1
  Related Headache | 100 | 45 | 46
  Any Muscle aches | 129 | 31 | 38
  Grade 3 Muscle aches | 6 | 0 | 0
  Related Muscle aches | 125 | 28 | 36
  Any Shivering | 95 | 19 | 26
  Grade 3 Shivering | 10 | 1 | 1
  Related Shivering | 94 | 17 | 22

5. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs).
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: During the 30-day (Days 0-29) follow-up period after vaccination
Population: The analysis was based on the Total Vaccinated Cohort which included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | GSK1247446A-AS03 Group | GSK1247446A Group | Fluarix Group
Number analyzed (Participants) | 407 | 406 | 407
Subjects
  Subjects with any AEs | 114 | 82 | 95
  Subjects with Grade 3 AEs | 13 | 11 | 16
  Subjects with related AEs | 43 | 19 | 19

6. Secondary Outcome: Number of Subjects With Any and Related Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity. Any = occurrence of any SAE regardless of intensity grade or relation to vaccination. Related = SAE assessed by the investigator as related to the vaccination.
Time Frame: During the entire study period (Day 0 to Day 180)
Population: The analysis was based on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | GSK1247446A-AS03 Group | GSK1247446A Group | Fluarix Group
Number analyzed (Participants) | 407 | 406 | 407
Subjects
  Subjects with any SAE(s) | 8 | 13 | 13
  Subjects with related SAE(s) | 2 | 1 | 0

ADVERSE EVENTS:
Time Frame: SAEs were collected during the entire study (Days 0-180). AEs were collected during the 30-day (Days 0-29) post-vaccination period. Solicited local/general symptoms were collected during the 7-day (Days 0-6) post-vaccination period.
Description: Non-serious AEs included solicited symptoms that were assessed on a subset of the Total Vaccinated Cohort, comprised of subjects who had symptom sheets completed.
Arm/Group | GSK1247446A-AS03 Group | GSK1247446A Group | Fluarix Group
Serious Adverse Events (participants affected / at risk) | 8/407 | 13/406 | 13/407
Other Adverse Events (participants affected / at risk) | 302/407 | 143/406 | 181/407
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1247446A-AS03 Group (N=407) | GSK1247446A Group (N=406) | Fluarix Group (N=407)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 — SAE reported from Day 0 to Day 30.
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0 — SAE reported from Day 0 to Day 30.
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 — SAE reported from Day 0 to Day 30.
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 — SAE reported from Day 0 to Day 30.
Grand mal convulsion (Nervous system disorders) | 0 | 1 | 0 — SAE reported from Day 0 to Day 30.
Injection site erythema (General disorders) | 1 | 0 | 0 — SAE reported from Day 0 to Day 30.
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 — SAE reported from Day 0 to Day 30.
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 — SAE reported from Day 0 to Day 30.
Pyrexia (General disorders) | 1 | 0 | 0 — SAE reported from Day 0 to Day 30.
Cerebral infarction (Nervous system disorders) | 2 | 0 | 1 — SAE reported from Day 30 to Day 180.
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 — SAE reported from Day 30 to Day 180.
Cholecystitis (Hepatobiliary disorders) | 1 | 1 | 0 — SAE reported from Day 30 to Day 180.
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 — SAE reported from Day 30 to Day 180.
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 — SAE reported from Day 30 to Day 180.
Brain stem thrombosis (Nervous system disorders) | 1 | 0 | 0 — SAE reported from Day 30 to Day 180.
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 — SAE reported from Day 30 to Day 180.
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 — SAE reported from Day 30 to Day 180.
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1 — SAE reported from Day 30 to Day 180.
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 — SAE reported from Day 30 to Day 180.
Diverticulitis (Infections and infestations) | 0 | 1 | 0 — SAE reported from Day 30 to Day 180.
Drowning (General disorders) | 0 | 0 | 1 — SAE reported from Day 30 to Day 180.
Extrasystoles (Cardiac disorders) | 0 | 0 | 1 — SAE reported from Day 30 to Day 180.
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 — SAE reported from Day 30 to Day 180.
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1 — SAE reported from Day 30 to Day 180.
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1 | 0 — SAE reported from Day 30 to Day 180.
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0 — SAE reported from Day 30 to Day 180.
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 — SAE reported from Day 30 to Day 180.
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 — SAE reported from Day 30 to Day 180.
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 — SAE reported from Day 30 to Day 180.
Peptic ulcer (Gastrointestinal disorders) | 0 | 1 | 0 — SAE reported from Day 30 to Day 180.
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 — SAE reported from Day 30 to Day 180.
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 — SAE reported from Day 30 to Day 180.
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 — SAE reported from Day 30 to Day 180.
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 — SAE reported from Day 30 to Day 180.
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1 | 0 — SAE reported from Day 30 to Day 180.
Uterine neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 — SAE reported from Day 30 to Day 180.
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 — SAE reported from Day 30 to Day 180.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1247446A-AS03 Group (N=407) | GSK1247446A Group (N=406) | Fluarix Group (N=407)
Arthralgia (General disorders) | 80 | 17 | 21
Fatigue (General disorders) | 149 | 42 | 47
Fever (General disorders) | 21 | 4 | 2
Headache (General disorders) | 104 | 51 | 53
Muscle aches (General disorders) | 129 | 31 | 38
Shivering (General disorders) | 95 | 19 | 26
Ecchymosis (General disorders) | 28 | 20 | 19
Pain (General disorders) | 246 | 32 | 86
Redness (General disorders) | 95 | 50 | 65
Swelling (General disorders) | 84 | 8 | 50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.